CLINICAL TRIAL: NCT02354833
Title: Phenylephrine vs. Norepinephrine Infusion in Preventing Hypotension After Spinal Anesthesia for Cesarean Delivery
Brief Title: Phenylephrine vs. Norepinephrine Infusion After Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Manuel C. Vallejo MD , DMD, Chair; Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1406316590
Record Dates: First submitted 2015-01-20; First posted 2015-02-03 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Effects of; Anesthesia, in Labor and Delivery
Keywords: Hypotension; Cesarean Delivery; Phenylephrine; Spinal Anesthesia; Norepinephrine
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine (Experimental): A continuous phenylephrine infusion at 0.1 mcg/kg/min
  Interventions: Drug: Phenylephrine
- Norepinephrine (Experimental): A continuous norepinephrine infusion at 0.05 mcg/kg/min
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine
  Arms: Phenylephrine
Drug: Norepinephrine
  Other Names: Levophed
  Arms: Norepinephrine

SUMMARY:
The purpose of the study is to determine if a medication called phenylephrine, which helps to control blood pressure, is more effective as a continuous intravenous (IV) infusion compared to continuous IV norepinephrine in maintaining blood pressure during a spinal anesthetic for a cesarean delivery. Good blood pressure control has been shown to decrease nausea and vomiting during and after cesarean delivery under spinal anesthesia. For elective cesarean delivery, all participants will receive spinal anesthesia with a local anesthetic and morphine (provides long term pain control after cesarean delivery). This study plans to enroll 80 pregnant research subjects 18 years and above. Patients will be randomly assigned according to a computer generated system to be in one of two groups.

DETAILED DESCRIPTION:
This study will be a prospective, experimental, observational, randomized open label, active treatment controlled trial.

After written and informed consent are obtained, the study participants are randomly assigned using a computer generated table to 1 of 2 treatment groups prior to cesarean delivery.

Group A will consist of: A continuous phenylephrine infusion 0.1 mcg/kg/min to maintain systolic blood pressure (SBP) within 100-120% of baseline before the spinal.

Group B will consist of: A continuous norepinephrine infusion 0.05 mcg/kg/min to maintain systolic blood pressure (SBP) within 100-120% of baseline before the spinal.

Patients will be admitted to holding area. Baseline arterial blood pressure and heart rate will be measured in supine position, with left uterine displacement. Baseline blood pressure will be calculated by taking the mean of three consecutive SBP measurements taken 5 minutes apart. IV will be placed. Intravenous ondansetron 4 mg and up to 500 mL of Lactated Ringers solution administered prior to induction of spinal anesthesia.

The primary endpoint is the number of provider interventions needed to maintain the SBP within 100-120% of baseline for both groups. The secondary endpoint is nausea measured with each provider intervention after induction of spinal anesthesia, and immediately following delivery with 11 point verbal rating scale (0 = no nausea, 10 = worst possible nausea). Patients will also be instructed to report episodes of nausea at any other time during the study. Emesis will be recorded whenever present during the surgical procedure.

Hypertensive episodes (SBP greater than 120% of baseline) will be treated with cessation of infusion. Infusion will be restarted when SBP has decreased to below the upper limit of the target range (120% of baseline SBP). If the infusion must be stopped on three occasions, it will be discontinued permanently and the blood pressure maintained with phenylephrine boluses only.

Bradycardia (HR less than 50 BPM) will be treated with glycopyrrolate 0.4mg IV or ephedrine 5 mg - 10 mg IV bolus.

Study participants will receive a standard spinal anesthetic consisting of 0.75% hyperbaric bupivacaine (1.6 mL) plus preservative free morphine (0.2 mg) and fentanyl (20 mcg) at L3-4 or L4-5 interspace (the standard of care for spinal anesthesia at Ruby Memorial Hospital). Prior to surgical incision, the spinal sensory level will be tested to the bilateral T4 dermatomal level which is necessary for cesarean section under spinal anesthesia. The patients will be positioned supine with a wedge placed under the right hip to avoid aortocaval compression. Both the patient and the clinical research assistant (who will collect data) will not be blinded as to the administered phenylephrine infusion or norepinephrine infusion. The study will end when care is transferred to the labor and delivery room nurse.

Measured variables will include blood pressure (BP), the number and type of provider interventions for control of blood pressure (BP), heart rate (HR), cardiac output (CO) as measured by a noninvasive CO monitor, APGAR scores at 1 and 5 minutes, nausea and vomiting, and fetal cord blood analysis at delivery.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) Physical Status classification 1 and 2
* Pregnant women with singleton pregnancy
* Gestational age greater than 36 weeks
* Cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Use of cardiac medication or medication for blood pressure control
* Cardiovascular disease
* Multiple gestation
* Gestation diabetes requiring insulin
* History of postoperative nausea and vomiting
* Refusal to be in study
* Gastric bypass surgery
* History of chronic opioid use (chronic pain syndrome)
* Emergent caesarean delivery for maternal and/or fetal distress
* Eclampsia
* Progressive neurologic disease
* Infection at insertion site
* Allergy to local anesthetics, narcotics or other study medications.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Afolabi BB, Lesi FE. Regional versus general anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004350. doi: 10.1002/14651858.CD004350.pub3. PMID 23076903
- [Background] Djabatey EA, Barclay PM. Difficult and failed intubation in 3430 obstetric general anaesthetics. Anaesthesia. 2009 Nov;64(11):1168-71. doi: 10.1111/j.1365-2044.2009.06060.x. PMID 19825049
- [Background] Ohpasanon P, Chinachoti T, Sriswasdi P, Srichu S. Prospective study of hypotension after spinal anesthesia for cesarean section at Siriraj Hospital: incidence and risk factors, Part 2. J Med Assoc Thai. 2008 May;91(5):675-80. PMID 18672631
- [Background] Lin FQ, Qiu MT, Ding XX, Fu SK, Li Q. Ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean section: an updated meta-analysis. CNS Neurosci Ther. 2012 Jul;18(7):591-7. doi: 10.1111/j.1755-5949.2012.00345.x. PMID 22759268
- [Background] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Background] Stewart A, Fernando R, McDonald S, Hignett R, Jones T, Columb M. The dose-dependent effects of phenylephrine for elective cesarean delivery under spinal anesthesia. Anesth Analg. 2010 Nov;111(5):1230-7. doi: 10.1213/ANE.0b013e3181f2eae1. Epub 2010 Sep 14. PMID 20841418
- [Background] Allen TK, George RB, White WD, Muir HA, Habib AS. A double-blind, placebo-controlled trial of four fixed rate infusion regimens of phenylephrine for hemodynamic support during spinal anesthesia for cesarean delivery. Anesth Analg. 2010 Nov;111(5):1221-9. doi: 10.1213/ANE.0b013e3181e1db21. Epub 2010 May 21. PMID 20495139
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Comparison of phenylephrine infusion regimens for maintaining maternal blood pressure during spinal anaesthesia for Caesarean section. Br J Anaesth. 2004 Apr;92(4):469-74. doi: 10.1093/bja/aeh088. Epub 2004 Feb 20. PMID 14977792
- [Background] Doherty A, Ohashi Y, Downey K, Carvalho JC. Phenylephrine infusion versus bolus regimens during cesarean delivery under spinal anesthesia: a double-blind randomized clinical trial to assess hemodynamic changes. Anesth Analg. 2012 Dec;115(6):1343-50. doi: 10.1213/ANE.0b013e31826ac3db. Epub 2012 Sep 25. PMID 23011562

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenylephrine: A continuous phenylephrine infusion at 0.1 mcg/kg/min
  Phenylephrine
- Norepinephrine: A continuous norepinephrine infusion at 0.05 mcg/kg/min
  Norepinephrine
Period: Overall Study
Arm/Group | Phenylephrine | Norepinephrine
Started | 38 | 43
Completed | 38 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We conducted a prospective, observational, randomized, open labeled trial on parturient scheduled for elective cesarean delivery under spinal anesthesia.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Norepinephrine | Total
Number analyzed (Participants) | 38 | 43 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 43 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.6) | 31.2 (6.8) | 30.15 (6.2)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 43 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Rescue Boluses to Maintain SBP
Description: Number of rescue boluses to maintain the SBP within 100-120% of baseline
Time Frame: At time of surgery, up to 2 hours
Measure: Number; unit: rescue boluses
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 38 | 43
rescue boluses | 25 | 21
Statistical Analysis 1: Comparison: Phenylephrine vs Norepinephrine; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

2. Secondary Outcome: Percentage of Participants Experiencing Both Nausea and Emesis
Time Frame: At time of surgery, up to 2 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phenylephrine; Norepinephrine: Cardiac Output as recorded by a non-invasive hemodynamic monitor
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 38 | 43
percentage of participants
  Percentage of participants with Nausea | 63.2 [47.9 to 78.5] | 51.2 [36.3 to 66.1]
  Percentage of participants with Emesis | 26.3 [12.3 to 40.3] | 16.3 [5.3 to 27.3]
Statistical Analysis 1: Comparison: Phenylephrine vs Norepinephrine; This analysis is comparing the percentage of participants with Nausea; Test type: Superiority or Other; p = 0.28, Chi-squared
Statistical Analysis 2: Comparison: Phenylephrine vs Norepinephrine; This analysis is comparing the percentage of participants with Emesis; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Primary Outcome: Median Total Rescue Bolus Dose of Ephedrine (mg) to Maintain SBP
Time Frame: At time of surgery, up to 2 hours
Measure: Median (Full Range); unit: mg
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 38 | 43
mg | 0 [0 to 85] | 0 [0 to 30]
Statistical Analysis 1: Comparison: Phenylephrine vs Norepinephrine; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Median Total Rescue Bolus Dose of Phenylephrine (mcg) to Maintain SBP
Time Frame: At time of surgery, up to 2 hours
Measure: Median (Full Range); unit: mcg
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 38 | 43
mcg | 50 [0 to 1000] | 100 [0 to 700]
Statistical Analysis 1: Comparison: Phenylephrine vs Norepinephrine; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Phenylephrine; Norepinephrine: Hypotension requiring a rescue bolus
Arm/Group | Phenylephrine | Norepinephrine
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/43
Other Adverse Events (participants affected / at risk) | 24/38 | 22/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenylephrine (N=38) | Norepinephrine (N=43)
Nausea (Gastrointestinal disorders) | 24 (24) | 22 (22)

LIMITATIONS AND CAVEATS:
38 subjects were enrolled in the phenylephrine group and none excluded. 47 subjects were enrolled in the norepinephrine group; 4 patients excluded (2 patients due to monitoring equipment failure, and 2 patients due to emergency cesarean deliveries).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes